CLINICAL TRIAL: NCT05814523
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Intravenous Ganaxolone Added to Standard of Care in Refractory Status Epilepticus
Brief Title: To Evaluate the Efficacy, Safety, and Tolerability of Intravenous Ganaxolone Added to Standard of Care in Refractory Status Epilepticus (RSE)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-SE-3004
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Refractory Status Epilepticus
Keywords: Refractory status epilepticus; Ganaxolone; Antiepileptic drug; Standard of care
MeSH Terms: conditions — Status Epilepticus | interventions — ganaxolone; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ganaxolone IV solution + SOC IV AED (Experimental)
  Interventions: Drug: Ganaxolone; Drug: Standard of care
- Placebo IV solution + SOC IV AED (Experimental)
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Ganaxolone — Ganaxolone will be administered as IV solution.
  Arms: Ganaxolone IV solution + SOC IV AED
Drug: Placebo — Placebo will be administered as IV solution.
  Arms: Placebo IV solution + SOC IV AED
Drug: Standard of care — A non-anesthetic medication not previously used for treatment of SE within the current episode and will be administered at a dose sufficient for the termination of SE according to investigator judgment.

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study that will evaluate the efficacy, safety, and tolerability of intravenous (IV) ganaxolone versus placebo co-administered with IV antiepileptic drug (AED) according to standard of care for the treatment of RSE. Approximately 70 participants will be randomized in a 1:1 ratio to receive ganaxolone IV solution or placebo IV solution along with standard of care (SOC) IV AED.

ELIGIBILITY:
Inclusion Criteria:

1. Participant, participant's parent, guardian, or LAR must provide signed informed consent/assent, and once capable (per institution guidelines), there must be documentation of consent/assent by the participant demonstrating they are willing and aware of the investigational nature of the study and related procedures. Where allowed by law, where the participant lacks the capacity to make informed decisions regarding his/her medical treatment options, the treating clinician may follow their deferred consenting practices. The clinician will make the final decision based on the best interests of the participant.
2. Male or females 18 years of age and older at the time of the first dose of IP.
3. SE warranting imminent progression of treatment meeting the following criteria:

   a) A diagnosis of SE, warranting imminent progression of treatment for seizure control, with or without prominent motor features based on clinical and EEG findings:

   i. Diagnosis is established by:
   * For SE with prominent motor features: Clinical and EEG seizure activity indicative of convulsive, myoclonic, or focal motor SE.
   * For SE without prominent motor features (nonconvulsive SE): Appropriate clinical features and an EEG indicative of non-convulsive status epilepticus (NCSE).

   ii. For any type of SE:
   * At least 6 minutes of cumulative seizure activity over a 30-minute period within the hour before IP initiation, AND Seizure activity during the 30 minutes immediately prior to IP initiation.
4. Participants must have received a benzodiazepine and at least 1 of the following IV AEDs for treatment of the current episode of SE administered at an adequate dose and for a sufficient duration, in the judgement of the investigator, to demonstrate efficacy. The benzodiazepine and at least 1 of the IV AEDs must have been administered at a dose that would be expected to be effective for the termination of the current episode of SE.

   * IV Fosphenytoin/phenytoin,
   * IV Valproic acid,
   * IV Levetiracetam,
   * IV Lacosamide,
   * IV Brivaracetam, or
   * IV Phenobarbital.
5. Body mass index (BMI) < 40 or, if BMI is not able to be calculated at screening, participant is assessed by investigator as not morbidly obese.

Exclusion Criteria:

1. Life expectancy of less than 24 hours.
2. Anoxic brain injury or an uncorrected, rapidly reversable metabolic condition as the primary cause of SE (eg, hypoglycemia < 50 milligrams per deciliter [mg/dL] or hyperglycemia > 400 mg/dL).
3. Participants who have received high-dose IV anesthetics (eg, midazolam, propofol, thiopental, or pentobarbital) during the current episode of SE for more than 18 hours, or who continue to have clinical or electrographic evidence of persistent seizures while receiving high-dose IV anesthetics.
4. Clinical condition or advance directive that would NOT permit admission to the ICU or use of IV anesthesia.
5. Participants known or suspected to be pregnant
6. Participants with known allergy or sensitivity to progesterone or allopregnanolone medications/supplements
7. Receiving a concomitant IV product containing Captisol.
8. Known or suspected hepatic insufficiency or hepatic failure leading to impaired synthetic liver function.
9. Known or suspected stage 3B (moderate to severe; estimated glomerular filtration rate [eGFR] 44-30 milliliters per minute per 1.73-meter square [mL/min/1.73m^2]), stage 4 (severe; eGFR 29-15 mL/min/1.73m^2), or stage 5 (kidney failure; eGFR < 15 mL/min/1.73m^2 or dialysis) kidney disease.
10. Use of an investigational product for which less than 30 days or 5 half-lives have elapsed from the final product administration. Participation in a non-interventional clinical study does not exclude eligibility.
11. Known or suspected history or evidence of a medical condition that, in the investigator's judgment, would expose a participant to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who will report cessation of SE within 30 minutes of investigational product (IP) initiation of at least 30 minutes duration | Up to 30 minutes
  Status epilepticus cessation will be determined by the investigator based on clinical and electroencephalography (EEG) features
Percentage of participants who will report no escalation of treatment for persistent or recurrent SE within 36 hours of IP initiation | Up to 36 hours

SECONDARY OUTCOMES:
Percentage of participants who will report cessation of SE within 30 minutes of IP initiation of at least 30 minutes duration | Up to 30 minutes
Percentage of participants who will report no escalation of treatment for persistent or recurrent SE within 72 hours of IP initiation | Up to 72 hours
Time to SE cessation | Up to 72 hours
Percentage of participants having cessation of SE within 30 minutes of IP initiation of at least 30 minutes duration without escalation of treatment | Up to 30 minutes
Percentage of participants reporting no escalation of treatment for persistent or recurrent SE within 36 hours of IP initiation | Up to 36 hours
Percentage of participants reporting no escalation of treatment for persistent or recurrent SE within 72 hours of IP initiation | Up to 72 hours
Change from Baseline in Modified Rankin Scale (mRS) at the time of hospital discharge | Baseline and Up to Day 31
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death where 0 - No symptoms; 1=No significant disability. Able to carry out all usual activities, despite some symptoms; 2=Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3=Moderate disability. Requires some help, but able to walk unassisted; 4=Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5=Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6=Dead. Higher scores will indicate high degree of disability.
Change from Baseline in level of responsiveness as assessed by the Full Outline of UnResponsiveness (FOUR) Score scale | Baseline and at 24, 36 and 72 hours
  The FOUR Score is a 17-point scale (with potential scores ranging from 0 - 16). Decreasing FOUR Score is associated with worsening level of consciousness. The FOUR coma scale includes 4 parameters with a minimum score of 0 and a maximum score of "4" for each of them: eye reactions (eye opening and tracking), motor responses (pain response and simple commands), stem reflexes (pupillary, corneal and cough) and respiratory patterns (respiratory rhythm and respiratory attempts in patients on a ventilator). The points are summed up, their sum is estimated. The interpretation of results will be as 15 to 16 score: clear consciousness; Less than 15: Impairment of consciousness; from 4 to 8: Coma and 0-4: Death. Lower the score, the greater the coma gravity.
Change from Baseline in level of sedation/ agitation as assessed by Richmond Agitation and Sedation Scale (RASS) | Baseline and at 24, 36 and 72 hours
  The RASS is a medical scale used to measure the agitation or sedation level. It is a 10-point scale that ranges from -5 to +4 with -5=unarousable and +4=combative. Zero means the patient is alert and calm. higher scores indicate more agitation.
Percentage of participants with mRS > 3 at the time of hospital discharge | Up to 122 hours
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death where 0 - No symptoms; 1=No significant disability. Able to carry out all usual activities, despite some symptoms. 2=Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3=Moderate disability. Requires some help, but able to walk unassisted. 4=Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5=Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6=Dead. Higher scores will indicate high degree of disability.
Change from Baseline in Clinical Global Impression-Improvement (CGI-I) following IP initiation and at hospital discharge | Baseline and at 24, 36, and 72 hours
  The CGI-I is a 7-point Likert scale that the parent(s)/caregiver(s)/legally authorized representative (LAR)(s) and clinician uses to rate the change in overall seizure control, behavior, safety, and tolerability after initiation of the IP relative to Baseline (prior to treatment with the IP). It was rated as: 1- "very much improved", 2- "much improved', 3- "minimally improved", 4- "no change", 5- "minimally worse", 6- "much worse", and 7- "very much worse". Higher scores indicated worse condition.
Number of hours on positive pressure ventilation attributable to the episode of SE or its treatment | Up to 4 Weeks
  Healthcare Utilization Questionnaires include the Hospitalization Questionnaire and the Positive Pressure Ventilation (PPV) and Intubation Questionnaire. The Hospitalization Questionnaire should be collected at hospital discharge or at final study visit/contact. The need for non-invasive or invasive ventilatory support within 24 hours prior to IP initiation and following IP initiation and within 48 hours following IP discontinuation should be collected as close as possible to the event.
Number of hours on positive pressure ventilation | Up to 4 Weeks
Length of stay (days) in intensive care unit (ICU) | Up to 4 Weeks
Length of stay (days) in hospital | Up to 4 Weeks
Percentage of participants requiring artificial ventilation after initiation of IP | Up to 122 hours
Percentage of participants not requiring IV anesthesia for SE treatment within 36 hours of IP initiation | Up to 36 hours
Percentage of participants not requiring IV anesthesia for SE treatment within 72 hours of IP initiation | Up to 72 hours
Percentage of participants not requiring IV anesthesia for SE treatment through the final study follow-up visit/contact | Up to 4 Weeks
Percentage of participants who do not develop super refractory status epilepticus (SRSE) through the final study follow-up visit/contact | Up to 4 Weeks
Change from Baseline in Euro Quality of Life (five-level EuroQoL five-dimensional [EQ-5D-5L]) score | Baseline and Up to 4 Weeks
  The EQ-5D-5L is the EuroQoL 5D-5L, a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the participant's health state. A positive score means quality of life improvement, a negative score, a worsening of quality of life. Higher scores indicate more problems.
Number of AEDs at discharge | Up to 122 hours
Percentage of participants requiring supplemental oxygen after initiation of IP | Up to 4 Weeks

CONTACTS AND LOCATIONS:
Locations (52):
- Austria (5):
  - Medical University of Innsbruck, Innsbruck
  - Kepler University Hospital, Linz
  - Kepler Universitätsklinikum GmbH, Linz
  - Paracelsus Medical University Salzburg, Christian Doppler University Hospital, Department of Neurology, Salzburg
  - Medical University Vienna, Vienna
- Belgium (3):
  - Hôpital Universitaire de Bruxelles - Hôpital Erasme, Brussels
  - UZA University Hospital Antwerpen, Edegem
  - University Hospitals Leuven, Leuven
- Croatia (2):
  - Dubrava University Hospital, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - Mazaryk University, Brno,The First Department of Neurology, Brno
  - University Hospital Ostrava, Ostrava
  - Motol University Hospital, Prague
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- France (4):
  - Hopital R. Salengro, Lille
  - Hospices Civils de Lyon, Lyon
  - CHRU Nancy, Nancy
  - Chu de Toulouse, Toulouse
- Germany (4):
  - University of Osnabruck, Dep of Neurology, Osnabrück, Osnabrück, Osnabruck
  - Universitätsklinikum Erlangen, Erlangen
  - Epilepsy Center Hessen, Marburg
  - Universität- und Rehabilitationskliniken Ulm, RKU, Ulm
- National Institute of Clinical Neurosciences, Budapest, Hungary
- Israel (4):
  - Soroka Medical Center, Beersheba, Beer-Sheva
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Tel Aviv
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Azienda Ospedaliero Universitaria Caregg, Florence
  - Università Cattolica del Sacro Cuore, Milan
  - Azienda Ospedaliera Universitaria di Modena, Modena
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Poland (6):
  - Oddział Neurologii z Pododdziałem Udarowym Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Katowice-Ochojec
  - Oddzial Kliniczny Neurologii, Szpital Uniwersytecki w Krakowie, Krakow, Krakow
  - Uniwersyteckie Centrum Kliniczne im. prof. K. Gibińskiego w Katowicach, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanisława Szyszko Śląskiego Uniwersytetu, Katowice
  - Samodzielny Publiczny Szpital Kliniczny, Lublin
  - WSS im Gromkowskiego, Wroclaw
- Slovakia (4):
  - II. Neurologická klinika SZU Fakultná nemocnica s poliklinikou F. D. Roosevelta Banská Bystrica, Banská Bystrica
  - SlovakiaNeurologická klinika SZU a UNB Nemocnica Ružinov Univerzitná nemocnica Bratislava, Bratislava
  - Neurologické oddelenie Nemocnica Agel Levoča a.s., Levoča
  - Neurologické oddelenie Fakultná nemocnica, Trnava
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Santa Creu i Sant Pau, Institut de Recerca Biomedica Sant Pau, Barcelona
  - Hospital Clinico San Carlos Madrid., Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
- United Kingdom (3):
  - Cardiff and Vale UHB, Cardiff
  - King's College Hospital, Department of Neurology, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No